CLINICAL TRIAL: NCT03996473
Title: An Open-label, Multicenter, Phase 1/2 Study of Radium-223 Dichloride in Combination With Pembrolizumab in Participants With Stage IV Non-small Cell Lung Cancer
Brief Title: Study to Test the Safety and How Radium-223 Dichloride an Alpha Particle-emitting Radioactive Agent Works in Combination With Pembrolizumab an Immune Checkpoint Inhibitor in Patients With Stage IV Non-small Cell Lung Cancer With Bone Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: LPLV reached on 30Jan2023. Study was closed early for feasibility reasons related to enrollment of first line IO naïve patients. Safety data is consistent with the known safety profile of both drugs and no new safety issues have been observed
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19781; 2018-003704-39 (EudraCT Number)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — radium Ra 223 dichloride; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Radium-223+Pembrolizumab (Experimental): Participants received radium-223 dichloride at 55 kBq/kg every 6 weeks in combination with pembrolizumab every 3 weeks.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY 88-8223); Drug: Pembrolizumab
- Phase 2 Cohort 1: Radium-223+Pembrolizumab (Experimental): Participants was planned to receive radium-223 dichloride at the maximum tolerated dose (MTD) to be determined in the Phase 1 part every 6 weeks in combination with 200 mg pembrolizumab every 3 weeks.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY 88-8223); Drug: Pembrolizumab
- Phase 2 Cohort 1: Pembrolizumab alone (Active Comparator): Participants was planned to receive 200 mg pembrolizumab every 3 weeks.
  Interventions: Drug: Pembrolizumab
- Phase 2 Cohort 2: Radium-223+Pembrolizumab (Experimental): Participants was planned to receive radium-223 dichloride at the MTD to be determined in the Phase 1 part every 6 weeks in combination with 200 mg pembrolizumab every 3 weeks.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY 88-8223); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY 88-8223) — 55 kBq/kg, intravenous (IV) injection, every 6 weeks for up to 6 administrations
  Arms: Phase 1: Radium-223+Pembrolizumab; Phase 2 Cohort 1: Radium-223+Pembrolizumab; Phase 2 Cohort 2: Radium-223+Pembrolizumab
Drug: Pembrolizumab — 200 mg, IV infusion, every 3 weeks for a maximum of up to 35 administrations

SUMMARY:
The purpose of the study was to determine the safety and test the efficacy of the combination of radium-223 dichloride and pembrolizumab in patients with stage IV non-small cell lung cancer (NSCLC) with bone metastases who either had not received any systemic therapy for their advanced disease or had progressed on prior immunologic checkpoint blockade with antibodies against the programmed cell death protein-(ligand) 1 (PD-1/PD-L1). In this study researchers wanted to measure tumor shrinkage in response to treatment and how long that shrinkage lasted and gathered information on safety. Pembrolizumab is an immunologic checkpoint blocker that promotes an immune response against the tumor. Radium-223 dichloride is an alpha particle-emitting radioactive agent which kills cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV NSCLC.

  * Phase 2 Cohort 1: No Epidermal Growth Factor Receptor (EGFR) / v-Raf murine sarcoma viral oncogene homolog B (BRAF) mutation or anaplastic lymphoma kinase (ALK)/ROS1 rearrangement. Treatment naïve (no prior systemic therapy) for their metastatic NSCLC.
  * Phase 2 Cohort 2: progression on prior treatment with an immune checkpoint inhibitor inhibitor. Prior treatment with platinum-based chemotherapy in combination or in sequence in line with local standard of care.
  * Phase 1 includes participants meeting either Cohort 1 or Cohort 2 criteria.
* Measurable disease per RECIST v1.1.
* At least 2 skeletal metastases.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Adequate bone marrow and organ function.
* Participants must be on a bone health agent (BHA) treatment, such as bisphosphonates or denosumab treatment unless such treatment is contraindicated or not recommended per investigator's judgement.

Exclusion Criteria:

* Previous or concurrent cancer within 3 years prior to enrollment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor. Phase 2 Cohort 2: was discontinued from that treatment due to a Grade 3 or higher immune-related AEs (irAEs).
* Known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Known history or presence of osteonecrosis of jaw.
* Ongoing infection >Grade 2 NCI-CTCAE v.5.0 requiring systemic therapy.
* Significant acute GI disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or ≥ NCI-CTCAE v.5.0 Grade 2 diarrhea of any etiology.
* History of osteoporotic fracture.
* Prior treatment with radium-223 dichloride or any therapeutic radiopharmaceutical.
* Prior radiotherapy within 21 days of planned start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Ccare San Marcos Cancer Center & Urology, San Marcos, California, United States
- UZ Gent, Ghent, Belgium
- Nederlands Kanker Instituut, Amsterdam, Netherlands
- Spain (3):
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 4 countries between 06 March 2020 (first participant first visit) and 30 January 2023 (last participant last visit).
Pre-assignment Details: Overall, 10 participants were screened. Of them, 2 participants were screen failures. 8 participants were assigned to study treatment, of which 7 received the study treatment and 1 participant never received the treatment in the Phase 1.
Groups:
- Radium-223 Dichloride + Pembrolizumab: Participants received radium-223 dichloride at 55 kBq/kg every 6 weeks in combination with pembrolizumab every 3 weeks.
Period: Treatment Assignment
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Started | 8
Completed | 0
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 6
Not completed — Study drug never administered | 1
Period: Active Follow-up
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1
Period: Long-term Follow-up
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Started | 6
Completed | 1
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): includes all participants who received at least 1 administration of study treatment.
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.7) [lower limit 10.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events in Phase 1
Description: A treatment-emergent adverse event (TEAE) was any untoward medical occurrence in a participant, whether or not related to the treatment, arising or worsening after start of study treatment administration until the end of treatment visit (EoT visit, i.e. 30 [+7] days after last dose of study treatment). Severities of the TEAEs are summarized overall and by the maximum grade experienced by the participants for any TEAEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.0.
Time Frame: Up to 218 days
Population: Safety analysis set (SAF): included all participants who received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Participants
  Any TEAE | 7
  Any TEAE - Maximum Grade 1 | 0
  Any TEAE - Maximum Grade 2 | 3
  Any TEAE - Maximum Grade 3 | 2
  Any TEAE - Maximum Grade 4 | 0
  Any TEAE - Maximum Grade 5 | 2

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events in Phase 1
Description: A treatment-emergent serious adverse event (TESAE) was any untoward medical occurrence that resulting in death, initial or prolonged inpatient hospitalization, life-threatening, persistent disability/incapacity, congenital anomaly/birth defect, another medical important serious event as judged by the investigator arising or worsening after start of study treatment administration until 90 days after the cessation of study treatment for serious AE (regardless of causality) or until the end of treatment visit (EoT visit, i.e. 30 [+7] days after last dose of study treatment) visit if the participant initiated new anti-cancer therapy, whichever was earlier.
Time Frame: Up to 278 days
Population: Safety analysis set (SAF): included all participants who received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 2

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Phase 1
Description: Any of following toxicities (exceptions as in protocol) during DLT window was considered a DLT if assessed by investigator to be possibly, probably or definitely related to study treatment: 1.Grade 4 non-hematologic toxicity. 2.Grade 4 hematologic toxicity ≥7 days. 3.Any non-hematologic AE (excl. lab) ≥Grade 3. 4.Any Grade 3 non-hematologic lab value if clinically significant medical intervention required, or the abnormality led to hospitalization, or the abnormality persisted for >1 week. 5.Grade 3 abnormality in AST, ALT, or bilirubin without liver metastases at screening; The abnormality results in a Drug-induced Liver Injury. 6.Febrile neutropenia Grade 3 or 4. 7.Prolonged delay (>2 weeks) in initiating Cycle 2 of pembrolizumab due to treatment-related toxicity 8.Any treatment-related toxicity that caused the participant to discontinue treatment during Cycle 1 or 2. 9.Missing >25% of pembrolizumab doses as a result of drug-related AE(s) during the first cycle. 10.Grade 5 toxicity.
Time Frame: Within 6 weeks after the first administration of pembrolizumab
Population: DLT analysis set: included all the following participants: a. participants who experienced a DLT during the DLT observation window; b. participants who did not experience a DLT, and who were not dropouts. Dropouts were eligible participants who withdrew during the DLT observation window (within 6 weeks after the first administration of pembrolizumab) for reasons other than experiencing a DLT, and who did not complete both 1 dose of radium-223 dichloride and 2 cycles of pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 6
Participants | 0

4. Primary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 in Phase 2
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) during the course of the study. It was evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1). Complete Response (CR): Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions.
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Categorized by Best Tumor Responses Per RECIST v1.1 in Phase 1
Description: The tumor responses were evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1).
Time Frame: Up to 188 days
Population: Efficacy analysis set (EFF): included all participants who received at least 1 administration of planned dose of any study treatment in Phase 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Participants
  Stable disease (SD) | 1
  Progressive disease (PD) | 5
  Missing | 1

6. Secondary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 in Phase 1
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) during the course of the study. It was evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1). Complete Response (CR): Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions. Number of participants with best overall response of CR or PR before early termination of the study is reported in the table below while percentage of participants is auto-calculated by ClinicalTrials.gov database.
Time Frame: Up to 188 days
Population: Efficacy analysis set: included all participants who received at least 1 administration of planned dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 0

7. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1 in Phase 1
Description: DoR was defined as the time interval from the date of first response (CR or PR) to the date of disease progression or death, whichever comes first. It was evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1). Complete Response (CR): Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions.
Time Frame: Up to 188 days
Population: DoR was not analyzed due to no responder was reported before the study termination among the low number of participants. Tumor responses are reported in a separated outcome measure.
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 in Phase 1
Description: DCR was defined as the percentage of participants with CR or PR, or SD for at least 6 weeks during the course of the study. It was evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1). Complete Response (CR): Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions. Stable Disease (SD): Steady state of disease. Number of participants with best overall response of CR or PR or SD is reported below while percentage of participants is auto-calculated by ClinicalTrials.gov database.
Time Frame: Up to 188 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 1

9. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1 in Phase 2
Description: as for outcome 7
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 in Phase 2
Description: DCR was defined as the percentage of participants with CR or PR, or SD for at least 6 weeks during the course of the study. It was evaluated per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST V1.1). Complete Response (CR): Disappearance of all clinical and radiological evidence of tumor (both target and non-target). Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non target lesions and no appearance of new lesions. Stable Disease (SD): Steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, no unequivocal progression of existing non target lesions and no appearance of new lesions.
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Progression Free Survival (PFS) Per RECIST v1.1 in Phase 2
Description: Progression free survival (PFS) was defined as the time from start of any study treatment to the date of earliest radiological progression per RECIST 1.1 or death due to any cause, whichever occurs first. Participants who were alive and without progression at the time of database cut-off would be censored at the date of the last evaluable tumor assessment. RECIST: Response Evaluation Criteria in Solid Tumors
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Overall Survival (OS) in Phase 2
Description: Overall survival (OS) was defined as the time from start of any study treatment to the date of death due to any cause. Participants who were alive at the time of database cut-off would be censored at the last date known to be alive or the database cut-off date, whichever occurs first.
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events in Phase 2
Description: An treatment-emergent adverse event (TEAE) was any untoward medical occurrence in a participant, whether or not related to the treatment, arising or worsening after start of study treatment administration until the end of treatment visit (EoT visit, i.e. 30 [+7] days after last dose of study treatment). Severities of the TEAEs are summarized overall and by the maximum grade experienced by the participants for any TEAEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.0.
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events in Phase 2
Description: as for outcome 2
Time Frame: 0 day as Phase 2 never started due to the early termination of the study
Population: No participant started in Phase 2 part of the study prior to study termination
Arm/Group | Radium-223 Dichloride + Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment to 90 days after cessation of study treatment or 30 days after last dose of study treatment (EoT visit) if subject started new anti-cancer therapy (whichever was earlier) for serious TEAEs; or until EoT visit for other TEAEs, with a maximum of 278 days
Description: Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the entire study before the last contact (i.e. from signing ICF until the end of follow-up)
Groups:
- Radium-223 + Pembrolizumab: Subjects received radium-223 dichloride every 6 weeks for up to 6 administrations in combination with pembrolizumab every 3 weeks for up to 35 cycles.
Arm/Group | Radium-223 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 + Pembrolizumab (N=7)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 + Pembrolizumab (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Asthenia (General disorders) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight decreased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated early during the Phase 1 part of the study. This decision was based on strategic considerations also acknowledging the recruitment challenges for the first-line population. Due to the early termination, tumor responses were only listed, none of the efficacy outcome measures were actually analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 120 days from the time submitted to the sponsor for review. If a multicenter publication is not published within 18 months after completion of the study and database lock at all research sites or any earlier termination or abandonment of the study, PI shall have the right to publish and present the results.

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03996473/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03996473/SAP_001.pdf